CLINICAL TRIAL: NCT01346085
Title: A Multi-step Trial Towards Single Donor Islet Transplantation in Type 1 Diabetic Patients, Using Calcineurin Inhibitor-free Immunosuppression
Brief Title: Calcineurin Inhibitor (CNI)-Free Immunosuppressive Regimen in T1D Patients Receiving Islet Transplantation
Acronym: ECIT-1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ospedale San Raffaele (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Piemonti Lorenzo, Director Islet Transplantation Program, Ospedale San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECIT-1
Record Dates: First submitted 2011-04-29; First posted 2011-05-02 (Estimated); Results first posted 2014-05-09 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Type 1 Diabetes
Keywords: islet transplantation; brittle diabetes; type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Interleukin 1 Receptor Antagonist Protein; Sirolimus; thymoglobulin; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CNI-free single-group (Experimental)
  Interventions: Drug: CNI free immunosuppression

INTERVENTIONS:
Drug: CNI free immunosuppression — Immunosuppression consisted of: (i) pre-Tx rapamycin treatment (0.1 mg/kg/day) for at least 30 days; (ii) induction therapy with ATG (1.5 mg/kg/day for 4 days starting at day -1) and a steroid bolus (methyl-prednisolone 500 mg, day -1) plus low dose steroids (prednisone, 10 mg/day) and interleukin-1 (IL-1) receptor antagonist (100 mg/day) for 2 weeks (with ATG and steroid bolus administered only prior to the 1st islet infusion; (iii) maintenance with rapamycin (0.1 mg/kg/day) plus mycophenolate mofetil (2 g/day).
  Other Names: Kineret, Rapamune, Thymoglobulin, Myfortic

SUMMARY:
Our final objective is to develop an adoptive therapy with tolerogenic donor-specific Tr1 cells in T1D patients undergoing pancreatic islet transplantation (Tx). The achievement of this objective depends by the availability of an immunosuppressive treatment (IS) compatible with the survival, function, and expansion of the transferred Tr1 cells. For this purpose the investigators design a CNI-free single-group, phase 1-2 trial excluding the ATG or anti-CD25 induction therapy after the 1st islet infusion

DETAILED DESCRIPTION:
We designed the clinical trial as a single-arm, phase 1-2 trial conducted in two transplant centers (San Raffaele Scientific Institute, Milan, Italy; Cell Isolation and Transplantation Center, University of Geneva, Geneva, Switzerland) which used a common protocol for islet preparation, post-transplantation patient management and data collection. The trial is exploratory in nature and the target enrollment is 10 patients. The recruitment is competitive between the two centers and each patient is to receive at least 10,000 IE/kg. Up to three islet infusions are allowed per patients until insulin independence is reached, provided that partial islet function (i.e., fasting C-peptide ≥0.3 ng/mL) is maintained between infusions. We planned an individual follow-up of 3 years after the last islet infusion.

Patients with type 1 diabetes are eligible for this study. Major criteria for inclusion are: age 18-65 years; type 1 diabetes with onset <40 years of age; insulin treatment of at least 5 years at the time of enrollment; stimulated C-peptide in response to arginine <0.5 ng/ml; multiple (three or more) daily insulin injections or Continuous Subcutaneous Insulin Infusion; self-blood glucose monitoring ≥3 times/day; high glycemic instability and/or hypoglycemia unawareness; inability to consistently attain a glycated hemoglobin target of <7.5 % without severe hypoglycemia (defined as an hypoglycemic episode requiring the assistance by another person for its resolution) in the past 36 months despite medical management by a diabetes specialist. Major criteria for exclusion are: HbA1c >12%; BMI >30 kg/m2, or insulin requirement > 0.8 IU/kg/day; poorly controlled hypertension; untreated proliferative diabetic retinopathy; presence or history of macroalbuminuria (>300mg/g day) or estimated glomerular filtration rate <60 ml/min/1.73 m2 for females or <70 ml/min/1.73 m2 for males.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-65yr
* ability to provide written informed consent and comply with the study protocol procedures
* clinical history of type 1 diabetes with onset <40yr of age, on insulin for at least 5yr at the time of enrollment
* absent stimulated C-peptide (<0.5ng/ml) in response to arginine
* multiple (three or more) daily insulin injections or insulin pump therapy
* self blood glucose monitoring ≥3 times/day, supervised by a specialist physician
* high glycemic instability and hypoglycemia unawareness
* inability to consistently attain a HbA1c < 7.5 % target without experiencing severe hypoglycemia (assistance by another person) in the past 36 months despite appropriate medical management.

Exclusion Criteria:

* HbA1c >12%
* BMI >30 kg/m2, or insulin requirement of > 0.8 IU/kg/day;
* poorly controlled hypertension;
* untreated proliferative diabetic retinopathy;
* presence or history of macroalbuminuria (>300mg/g day) or measured glomerular filtration rate <60 ml/min/1.73 m2 for females and <70 ml/min/1.73 m2 for males
* for female participants: positive pregnancy test, presently breast-feeding, or unwilling to use effective contraceptive measures for the duration of the study and 3 months after discontinuation
* for male participants: intent to procreate during the duration of the study or within 3 months after discontinuation or unwillingness to use effective measures of contraception;
* any history of malignancy within the previous 5 years, except for completely resected squamous or basal cell carcinoma of the skin;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-10; Primary Completion 2009-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Piemonti, MD, Principal Investigator — Fondazione Centro San Raffaele del Monte Tabor; Thierry Berney, MD, Principal Investigator — Universitè de Geneve; Antonio Secchi, MD, Study Chair — Fondazione Centro San Raffaele del Monte Tabor; Paola Maffi, MD, Study Director — Cantro San Raffaele del Monte Tabor
Locations (2):
- IRCCS San Raffaele Scientific Institute, Milan, Italy
- Universitè de Geneve, Geneva, Switzerland

REFERENCES:
- [Background] Piemonti L, Maffi P, Monti L, Lampasona V, Perseghin G, Magistretti P, Secchi A, Bonifacio E. Beta cell function during rapamycin monotherapy in long-term type 1 diabetes. Diabetologia. 2011 Feb;54(2):433-9. doi: 10.1007/s00125-010-1959-6. Epub 2010 Nov 3. PMID 21046356
- [Result] Melzi R, Maffi P, Nano R, Sordi V, Mercalli A, Scavini M, Secchi A, Bonifacio E, Piemonti L. Rapamycin does not adversely affect intrahepatic islet engraftment in mice and improves early islet engraftment in humans. Islets. 2009 Jul-Aug;1(1):42-9. doi: 10.4161/isl.1.1.8881. PMID 21084848
- [Derived] Maffi P, Berney T, Nano R, Niclauss N, Bosco D, Melzi R, Mercalli A, Magistretti P, De Cobelli F, Battaglia M, Scavini M, Demuylder-Mischler S, Secchi A, Piemonti L. Calcineurin inhibitor-free immunosuppressive regimen in type 1 diabetes patients receiving islet transplantation: single-group phase 1/2 trial. Transplantation. 2014 Dec 27;98(12):1301-9. doi: 10.1097/TP.0000000000000396. PMID 25286053
- [Derived] Piemonti L, Everly MJ, Maffi P, Scavini M, Poli F, Nano R, Cardillo M, Melzi R, Mercalli A, Sordi V, Lampasona V, Espadas de Arias A, Scalamogna M, Bosi E, Bonifacio E, Secchi A, Terasaki PI. Alloantibody and autoantibody monitoring predicts islet transplantation outcome in human type 1 diabetes. Diabetes. 2013 May;62(5):1656-64. doi: 10.2337/db12-1258. Epub 2012 Dec 28. PMID 23274902

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CNI-free Single-group
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CNI-free Single-group
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (4.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Region of Enrollment [Number; unit: participants]
  Italy | 8
  Switzerland | 2

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Insulin Free Patients 3 Years After the Last Islet Infusion
Description: Insulin independence is defined as no need for exogenous insulin, with adequate glycemic control [i.e., glycated hemoglobin <7% (normal range 3.5 - 6.0%), fasting glucose levels not exceeding 140 mg/dL (7.8 mmol/L) more than three times per week and 2-hour postprandial levels not exceeding 180 mg/dL (10 mmol/L) more than four times per week].
Time Frame: 3 year
Measure: Number; unit: participants
Arm/Group | CNI-free Single-group
Number analyzed (Participants) | 10
participants | 4

2. Secondary Outcome: Insulin Independence With Adequate Glycemic Control Throughout Follow-up
Time Frame: up to 3 years
Measure: Number; unit: participants
Arm/Group | CNI-free Single-group
Number analyzed (Participants) | 10
participants | 4

3. Secondary Outcome: Glycated Hemoglobin Levels Throughout Follow-up
Time Frame: up to 3 years
Reporting Status: Not Posted

4. Secondary Outcome: Basal and Stimulated Blood C-peptide Levels in Response to Arginine Challenge Throughout Follow-up
Time Frame: up to 3 year
Reporting Status: Not Posted

5. Secondary Outcome: the Reduction in Insulin Requirement Compared to Baseline
Time Frame: up to 3 years
Reporting Status: Not Posted

6. Secondary Outcome: Severe Hypoglycemic Events Since Completion of Transplant
Time Frame: up to 3 years
Reporting Status: Not Posted

7. Secondary Outcome: Any Adverse Event Throughout Follow-up
Description: Among study participants there were no reports of death, post-transplantation lymphoproliferative disease, cancer, or opportunistic infections. There was no evidence of cytomegalovirus disease, infection or serological activation (CMV early antigens negative during the whole follow-up), nor of Epstein-Barr clinical and serological reactivation (all patients were antibodies anti EBV positive before transplant, as per the inclusion criteria).
Time Frame: up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 3 years after last islet infusion
Description: AEs were recorded according to the "Terminology Criteria for Adverse Events (TCAE) In Trials of Adult Pancreatic Islet Transplantation, Version 4.1 (16 July 2008)" (http://www.isletstudy.org/CITDocs/CIT-TCAE%20V4.pdf).
Arm/Group | CNI-free Single-group
Serious Adverse Events (participants affected / at risk) | 8/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CNI-free Single-group (N=10)
Leucopenia (Immune system disorders) | 8 (8)
Neutropenia (Immune system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Gastrointestinal conditions (Gastrointestinal disorders) | 2 (2)
ATG reaction during third infusion (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CNI-free Single-group (N=10)
Hemorrhage/bleeding from percutaneous transhepatic portal access (Surgical and medical procedures) | 5 (6) — Procedure-related adverse events included hemorrhage/bleeding from percutaneous transhepatic portal access in 6 of 20 islet infusions (30%)
Transient liver enzyme increase exceeding 5 times the baseline level (Gastrointestinal disorders) | 2 (2) — Transient liver enzyme increase was always observed after each islet infusion, and in 2 out of 20 procedures (10%) the observed increase exceeded 5 times the baseline level
Leucopenia (Immune system disorders) | 2 (2)
Mouth ulcers (Gastrointestinal disorders) | 9 (9)
Neutropenia (Immune system disorders) | 7 (7)
Anemia (Blood and lymphatic system disorders) | 6 (6)
Acne or rash (Skin and subcutaneous tissue disorders) | 6 (6)
Hyperlipemia (Metabolism and nutrition disorders) | 4 (4)
Gastrointestinal conditions (Gastrointestinal disorders) | 1 (1)
Fungal infection (Infections and infestations) | 3 (3) — Oral or vaginal candidiasis
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Peripheral edema (Skin and subcutaneous tissue disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Lower urinary tract infection (Infections and infestations) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes